CLINICAL TRIAL: NCT07259096
Title: Comparison of Knowledge Levels of Regular Conditioning Workers With and Without a History of Injury Regarding Sports Anxiety, Sports Injury Anxiety, and Factors Causing Injury in Sports
Brief Title: Comparison of Sports Anxiety, Sports Injury Anxiety, and Knowledge Levels Regarding Factors Causing Sports Injury in Individuals Who Regularly Engage in Conditioning Work With and Without a History of Injury
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Ilayda Dilan Isik, Msc, Physiotherapist, Istanbul Saglik Bilimleri University
Other Study IDs: AnkaraSBU2
Record Dates: First submitted 2025-11-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: People Who Do Regular Conditioning Work
Keywords: Conditioning Work; Sports Anxiety; Sports Injury Anxiety; Factors Causing Sports Injury; History of Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With a History of Injury
- Without a History of Injury

SUMMARY:
Anxiety, or anxiety disorder, is a common occurrence today. Studies have proven that sports have a high potential for stress and anxiety. Among the reasons for its prevalence in athletes are performance pressure, public scrutiny, dissatisfaction with athletic careers, injuries, and harassment and abuse in sports. Anxiety can negatively impact performance and competition results. However, the relationship between anxiety and performance has not been fully established. Studies on the relationship between anxiety and injury in athletes are also increasing. However, studies examining injury history and sports anxiety levels in individuals who regularly perform conditioning exercises are lacking.

Based on our literature review, our study will ask individuals who regularly engage in conditioning training about their injury history. Participants will be divided into two groups: those with and those without injuries. The two groups will be compared in terms of their sports anxiety and fear of injury, and their knowledge of the factors that contribute to injuries in sports will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Must have been doing regular conditioning exercises for at least 6 months
* Must be between 18-45 years of age

Exclusion Criteria:

* Being a professional athlete
* Having a neurological problem

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People who do regular conditioning work
Sampling Method: Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Sports Injury Anxiety | Last 3 months
  The assessment will be conducted using the Sport Anxiety Scale-2 (SAS-2). The questionnaire consists of a total of 15 items. Each item is scored between 1 and 4. An increase in the total score is interpreted as an increase in sport anxiety.
Sports Anxiety | Last 3 months
  The assessment will be conducted using the Sport Injury Anxiety Scale (SIAS). The scale was developed in 2016. The scale consists of 21 items, and each item is scored between 1 and 5. An increase in the score leads to the conclusion that the individual's sport injury anxiety has increased.
Level of Knowledge Regarding Factors Causing Injuries in Sports | Last 3 months
  The assessment will be conducted using the Factors Causing Sport Injury Scale (FCSIS).
  The scale was developed in 2023, and it is valid and reliable. An increase in the score obtained from the scale leads to the conclusion that the athlete is less affected by the related dimension of the factors causing injury.
  It consists of a total of 26 items, and each item is scored between 1 and 5. The questionnaire consists of 4 sub-dimensions. These are: personal factors, psychological factors, environmental factors, and coach-related factors.

CONTACTS AND LOCATIONS:
Locations (1):
- GYM Center, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Caz, Ç., Kayhan, R.F., & Bardakçı S. (2019). Adaptation of the sport injury anxiety scale to Turkish: Validity and reliability study. Turkish Journal of Sports Medicine, 54(1), 52-63. doi: 10.5152/tjsm.2019.116
- [Background] Akman, H., Yetkin Tekin, A., Tekin, A. (2025). Sport Anxiety Scale-2: Reliability and validity study in Turkish wrestlers. Turk J Sports Med. https://doi.org/10.47447/tjsm.0864
- [Background] Kolt GS, Kirkby RJ. Injury, anxiety, and mood in competitive gymnasts. Percept Mot Skills. 1994 Jun;78(3 Pt 1):955-62. doi: 10.1177/003151259407800351. PMID 8084718
- [Background] Reardon CL, Gorczynski P, Hainline B, Hitchcock M, Rice S. Anxiety Disorders in Athletes. Clin Sports Med. 2024 Jan;43(1):33-52. doi: 10.1016/j.csm.2023.06.002. Epub 2023 Jul 11. PMID 37949513
- [Background] Ford JL, Ildefonso K, Jones ML, Arvinen-Barrow M. Sport-related anxiety: current insights. Open Access J Sports Med. 2017 Oct 27;8:205-212. doi: 10.2147/OAJSM.S125845. eCollection 2017. PMID 29138604